CLINICAL TRIAL: NCT02582281
Title: The Non Touch Technique for Intrauterine Device Insertion, a Single Blinded Randomized Control Trial
Brief Title: Non Touch Technique for IUD Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CU161020
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non touch technique (Experimental): the intrauterine device TCu 380A will be inserted in the conventional method as follows: First, insert the speculum and view the cervix. The position of the cervix will very often confirm if the uterus is anteverted or retroverted. Second, using the Allis forceps hold the back of a cotton-ball swab and dip it into a povidine-iodine disinfectant solution, or equivalent. Swab the cervix. Then cut the threads to the appropriate length and remove the speculum.
  This technique omits the sounding of the uterus which is considered a quintessential procedure before IUD insertion for which there is no one established piece of evidence.The IUD is checked afterwards by transvaginal ultrasound.
  Interventions: Device: intrauterine device TCu 380A
- Traditional IUD insertion (Experimental): the intrauterine device TCu 380A will be inserted in the conventional method, and checked afterwards by transvaginal ultrasound.
  Interventions: Device: intrauterine device TCu 380A

INTERVENTIONS:
Device: intrauterine device TCu 380A
  Other Names: TCu 380A

SUMMARY:
The non touch technique is a modification of the traditional intrauterine device insertion technique. It abolishes the use of Allis and uterine sounding.

ELIGIBILITY:
Inclusion Criteria:

* Females desiring contraception with the use of IUD

Exclusion Criteria:

* Are pregnant or think they may be pregnant
* Septic pregnancy or abortion
* Have unexplained abnormal vaginal bleeding
* Have untreated cervical cancer
* Have malignant gestational trophoblastic disease
* Have uterine cancer
* Have uterine abnormalities
* Have or may have had a pelvic infection within the past three months
* Have or may have any sexually transmitted disease
* Have pelvic tuberculosis
* Are postpartum between 48 hours and 4 weeks
* Have benign gestational trophoblastic disease
* Have ovarian cancer
* Have AIDS (unless clinically well on anti-retroviral therapy)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
degree of pain during IUD insertion | 5 months
  Pain will be assessed by the use of visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt